CLINICAL TRIAL: NCT01651117
Title: Using Peer Mentors to Support PACT Team Efforts to Improve Diabetes Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 12-407
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; Mentors; Glucose control; Hemoglobin A, Glycosylated; Randomized Controlled Trial; Veterans
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual Care (No Intervention): Enrolled in two different time frames. No interventions will be provided to this arm. They will complete planned surveys, and blood draws (baseline, 6 months, and 12 months).
- Peer Mentoring (Experimental): Participants in this arm will be mentored for 6 months by a veteran who was once in poor control but is now in good control. They will then be further randomized to either becoming a mentor for 6 months or having no other additional active intervention. All participants in this arm will be evaluated in person at baseline, 6 months, 12 months, and 18 months.
  Interventions: Behavioral: Peer Mentoring
- Peer Mentoring FFM (from former mentee) (Experimental): Participants in this arm will be mentored by the former mentee for 6 months and will be followed in person for an additional 6 months after the completion of the active intervention.
  Interventions: Behavioral: Peer Mentoring

INTERVENTIONS:
Behavioral: Peer Mentoring — Patients will receive peer mentoring.
  Arms: Peer Mentoring; Peer Mentoring FFM (from former mentee)

SUMMARY:
The purpose of this study is to test the effectiveness of a peer mentor model in a mixed race population of poorly controlled diabetic Veterans. Also, the study aims to assess the effects of becoming a mentor on those who originally were mentees. It is expected that participants in the peer mentoring arms (Arm 2 and 3) will have improved glucose control regardless of race or ethnicity at the end of the intervention.

DETAILED DESCRIPTION:
The primary objectives of this study are: (1) test the long-term effectiveness of a peer mentor model on improving glucose control, blood pressure, LDL levels, diabetes mellitus quality of life, and depression scores in a mixed race population of poorly controlled diabetic Veterans; (2) test the effectiveness of using former peer mentees as peer mentors as a means of creating a self-sustaining program; and (3) and test the effects of becoming a mentor on those who were originally mentees given a growing literature that being a mentor is good for your health. Secondary objectives include: (1) in those randomized to being a mentee, explore mentor characteristics associated with improved HbA1c.

This study will be a prospective randomized controlled trial. Outcomes to be measured include glycosylated hemoglobin, blood pressure, direct LDL, diabetes quality of life and depression.

The trial has two phases. In phase one, patients with poorly controlled diabetes are randomized to usual care or receiving peer mentoring. In phase two, poorly controlled diabetics are randomized to usual care or receiving peer mentoring from former mentees. Former mentees from phase 1 are also randomized such that they will have a 50% chance of becoming a mentor.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* All participants must have a diagnosis of Type 2 diabetics.
* Diabetes began after age 30
* Mentees: Have an HbA1c > 8% on 2 different occasions in the course of 24 months, with at least one measure within 3 months of enrollment
* Mentors for Phase 1: Had an HbA1c of > 8% in the past 3 years and an HbA1c < (or equal to) 7.5% within 3 months of enrollment
* Mentors for Phase 2: Former mentee

Exclusion Criteria:

Exclusion Criteria:

* Does not speak English
* Unable to understand consents
* Severe speech impediment
* over the age of 75

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A. Long, MD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request of the PI

REFERENCES:
- [Derived] Long JA, Ganetsky VS, Canamucio A, Dicks TN, Heisler M, Marcus SC. Effect of Peer Mentors in Diabetes Self-management vs Usual Care on Outcomes in US Veterans With Type 2 Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2020 Sep 1;3(9):e2016369. doi: 10.1001/jamanetworkopen.2020.16369. PMID 32915236

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1 Usual Care: Poorly controlled diabetics randomized to no intervention will complete planned surveys, and blood draws (baseline, 6 months, and 12 months).
- Stage 1 Peer Mentoring: Poorly controlled diabetics randomized to intervention will be mentored for 6 months by a veteran who was once in poor control but is now in good control.
  For stage 2, they will then be further randomized to either becoming a mentor for 6 months or having no other additional active intervention. All participants in this arm will be evaluated in person at baseline, 6 months, 12 months, and 18 months.
- Stage 2 Usual Care: Poorly controlled diabetics randomized to stage 2 no intervention will complete planned surveys, and blood draws (baseline, 6 months, and 12 months).
- Stage 2 Peer Mentoring FFM (From Former Mentee): Poorly controlled diabetics randomized to stage 2 intervention will be mentored by the former mentee for 6 months and will be followed in person for an additional 6 months after the completion of the active intervention.
Period: Overall Study
Arm/Group | Stage 1 Usual Care | Stage 1 Peer Mentoring | Stage 2 Usual Care | Stage 2 Peer Mentoring FFM (From Former Mentee)
Started | 156 | 205 | 49 | 70
Completed | 154 | 202 | 47 | 68
Not Completed | 2 | 3 | 2 | 2
Not completed — Death | 2 | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1 Usual Care | Stage 1 Peer Mentoring | Stage 2 Usual Care | Stage 2 Peer Mentoring FFM (From Former Mentee) | Total
Number analyzed (Participants) | 154 | 202 | 47 | 68 | 471
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (7.4) | 59.6 (7.9) | 62.3 (6.8) | 62.3 (6.9) | 60.6 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 0 | 2 | 17
  Male | 146 | 195 | 47 | 66 | 454
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 4 | 1 | 27
  Not Hispanic or Latino | 143 | 191 | 43 | 67 | 444
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 40 | 50 | 9 | 20 | 119
  Black | 93 | 136 | 37 | 45 | 311
  Multiple Race | 2 | 5 | 0 | 3 | 10
  Other Race | 19 | 11 | 1 | 0 | 31
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 154 | 202 | 47 | 68 | 471
Baseline HbA1c [Mean (Standard Deviation); unit: percent] | 9.8 (1.6) | 9.3 (1.6) | 9.7 (2.0) | 9.2 (1.7) | 9.5 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glucose Control (Stage 1: Usual Care v. Peer Mentoring)
Description: Measured by change in HbA1c, adjusted for baseline HbA1c and patient random effects. HbA1c is measured as a percent. Values of the change variable (difference of 2 percentages) can be positive or negative. Negative change, which shows better outcome, occurs when the 6 month HBA1c is lower than the baseline HbA1c. (Change = final measure - initial measure)
Time Frame: Baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: percent
Groups:
- Stage 1 Usual Care: Poorly controlled diabetics randomized to no interventions will complete planned surveys, and blood draws (baseline, 6 months, and 12 months).
- Stage 1 Peer Mentoring: Poorly controlled diabetics randomized to intervention will be mentored for 6 months by a veteran who was once in poor control but is now in good control.
Arm/Group | Stage 1 Usual Care | Stage 1 Peer Mentoring
Number analyzed (Participants) | 154 | 202
percent | -0.1978 [-0.4567 to 0.0611] | -0.5246 [-0.7554 to -0.2939]
Statistical Analysis 1: Comparison: Stage 1 Usual Care vs Stage 1 Peer Mentoring; Test type: Equivalence — Mixed methods ANCOVA with patient random effects, to compare change in HbA1c from baseline to 6 months between treatment and control groups; p = 0.0611, Mixed Models Analysis — Subject random effect included because same model was used for analyses of 2 separate follow up periods (baseline to 6 month, and baseline to 12 month, reported separately); Multiple imputation used for intent-to-treat analysis; Mean Difference (Final Values) = -0.3268, 95% CI 2-sided [-0.6690 to 0.0154], Standard Error of Mean 0.1739 — Negative parameter estimate means decrease in HbA1c was greater for treatment group than for control group

2. Primary Outcome: Change in Glucose Control (Stage 2: Usual Care v. Mentees)
Description: as for outcome 1
Time Frame: Baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Stage 2 Usual Care | Stage 2 Peer Mentoring FFM (From Former Mentee)
Number analyzed (Participants) | 47 | 68
percent | -0.4587 [-1.0223 to 0.1049] | 0.0772 [-0.4159 to 0.5703]

3. Primary Outcome: Change in Glucose Control (Stage 2: Non-mentors v. Mentors)
Description: as for outcome 1
Time Frame: Baseline to 6 months
Population: After 6 month of Stage 1, patients who were randomized to receive mentoring in Stage 1 were further randomized to either become a mentor in Stage 2 (Stage 2 Mentor) or to not become a mentor in Stage 2 (Stage 2 Non-mentor). Note that only those who had a 6-month follow-up visits for Stage 1 could be randomized to Stage 2 (139 participants).
Measure: Mean (95% Confidence Interval); unit: percent
Groups:
- Stage 2 Non-mentor: Patients who received peer mentoring in stage 1 who were randomized to no further treatment.
- Stage 2 Mentor: Patients who received peer mentoring in stage 1 who were randomized to become mentors to poorly controlled diabetics.
Arm/Group | Stage 2 Non-mentor | Stage 2 Mentor
Number analyzed (Participants) | 69 | 70
percent | 0.3156 [-0.0733 to 0.7045] | 0.1449 [-0.2421 to 0.5319]

4. Secondary Outcome: Change in Direct LDL Blood Levels
Description: Measured by change in Direct LDL blood levels, adjusted for baseline LDL and patient random effect. LDL is measured as mg/dL. Values of the change variable (difference of 2 levels) can be positive or negative. Negative change, which shows better outcome, occurs when the 6 month LDL is lower than the baseline LDL. (Change = final measure - initial measure)
Time Frame: Baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Stage 1 Usual Care | Stage 1 Peer Mentoring
Number analyzed (Participants) | 154 | 202
mg/dL | -2.0793 [-6.5786 to 2.4199] | -4.3098 [-8.3135 to -0.3061]

5. Secondary Outcome: Change in Systolic Blood Pressure
Description: Measured by change in systolic Blood Pressure, adjusting for baseline blood pressure and patient random effect. Systolic BP is measured as mmHG. Values of the change variable (difference of 2 levels) can be positive or negative. Negative change, which shows better outcome, occurs when the 6 month BP is lower than the baseline BP. (Change = final measure - initial measure)
Time Frame: Baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: mmHG
Arm/Group | Stage 1 Usual Care | Stage 1 Peer Mentoring
Number analyzed (Participants) | 154 | 202
mmHG | -3.4477 [-6.2332 to -0.6623] | -0.8695 [-3.4789 to 1.7399]

6. Secondary Outcome: Change in Diabetes Quality of Life Score
Description: Change in Diabetes Distress Scale, adjusted for baseline score and patient random effects. The DDS score is calculated by averaging 2 5-point Likert scale questions, and ranges from 1 to 5, where lower means less distress. Values of the change variable can be positive or negative. Negative change, which shows better outcome, occurs when the 6 month DDS is lower than the baseline DDS. (Change = final measure - initial measure)
Time Frame: Baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stage 1 Usual Care | Stage 1 Peer Mentoring
Number analyzed (Participants) | 154 | 202
score on a scale | 0.0159 [-0.1443 to 0.1761] | -0.0371 [-0.2036 to 0.1294]

7. Secondary Outcome: Change in Depression Symptoms
Description: As measured by change in the Patient Health Questionnaire-2, adjusted for baseline score and patient random effects. The PHQ score is calculated by summing 2 4-point 0-3 Likert scale questions, and ranges from 0 to 6, with lower score indicating lower depression. Values of the change variable can be positive or negative. Negative change, which shows better outcome, occurs when the 6 month PHQ is lower than the baseline PHQ. (Change = final measure - initial measure)
Time Frame: Baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stage 1 Usual Care | Stage 1 Peer Mentoring
Number analyzed (Participants) | 154 | 202
score on a scale | -0.0502 [-0.2792 to 0.1788] | -0.0389 [-0.2561 to 0.1782]

8. Secondary Outcome: Change in Glucose Control
Description: Measured by change in HbA1c, adjusted for baseline HbA1c and patient random effects. HbA1c is measured as a percent. Values of the change variable (difference of 2 percentages) can be positive or negative. Negative change, which shows better outcome, occurs when the 12 month HBA1c is lower than the baseline HbA1c. (Change = final measure - initial measure)
Time Frame: Baseline to 12 months
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Stage 1 Usual Care | Stage 1 Peer Mentoring
Number analyzed (Participants) | 154 | 202
percent | -0.2643 [-0.5263 to -0.0024] | -0.2818 [-0.5311 to -0.0326]

9. Secondary Outcome: Change in Direct LDL Blood Levels
Description: Measured by change in Direct LDL blood levels, adjusted for baseline LDL and patient random effect. LDL is measured as mg/dL. Values of the change variable (difference of 2 levels) can be positive or negative. Negative change, which shows better outcome, occurs when the 12 month LDL is lower than the baseline LDL. (Change = final measure - initial measure)
Time Frame: Baseline to 12 months
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Stage 1 Usual Care | Stage 1 Peer Mentoring
Number analyzed (Participants) | 154 | 202
mg/dL | -7.1706 [-11.7706 to -2.5705] | -7.8594 [-12.4047 to -3.3140]

10. Secondary Outcome: Change in Systolic Blood Pressure
Description: Measured by change in systolic Blood Pressure, adjusting for baseline blood pressure and patient random effect. Systolic BP is measured as mmHG. Values of the change variable (difference of 2 levels) can be positive or negative. Negative change, which shows better outcome, occurs when the 12 month BP is lower than the baseline BP. (Change = final measure - initial measure)
Time Frame: Baseline to 12 months
Measure: Mean (95% Confidence Interval); unit: mmHG
Arm/Group | Stage 1 Usual Care | Stage 1 Peer Mentoring
Number analyzed (Participants) | 154 | 202
mmHG | -3.7548 [-6.5977 to -0.9118] | -2.3274 [-4.9242 to 0.2695]

11. Secondary Outcome: Change in Diabetes Quality of Life
Description: Change in Diabetes Distress Scale, adjusted for baseline score and patient random effects. The DDS score is calculated by averaging 2 5-point Likert scale questions, and ranges from 1 to 5, where lower means less distress. Values of the change variable can be positive or negative. Negative change, which shows better outcome, occurs when the 12 month DDS is lower than the baseline DDS. (Change = final measure - initial measure)
Time Frame: Baseline to 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stage 1 Usual Care | Stage 1 Peer Mentoring
Number analyzed (Participants) | 154 | 202
score on a scale | -0.1213 [-0.2869 to 0.0414] | -0.1812 [-0.3445 to -0.0179]

12. Secondary Outcome: Change in Depression Symptoms
Description: As measured by change in the Patient Health Questionnaire-2, adjusted for baseline score and patient random effects. The PHQ score is calculated by summing 2 4-point 0-3 Likert scale questions, and ranges from 0 to 6, with lower score indicating lower depression. Values of the change variable can be positive or negative. Negative change, which shows better outcome, occurs when the 12 month PHQ is lower than the baseline PHQ. (Change = final measure - initial measure)
Time Frame: Baseline to 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stage 1 Usual Care | Stage 1 Peer Mentoring
Number analyzed (Participants) | 154 | 202
score on a scale | -0.1168 [-0.3472 to 0.1135] | -0.1736 [-0.3880 to 0.0407]

13. Secondary Outcome: Change in Direct LDL Blood Levels (Stage 2: Usual Care v. Mentees)
Description: as for outcome 4
Time Frame: Baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Stage 2 Usual Care | Stage 2 Peer Mentoring FFM (From Former Mentee)
Number analyzed (Participants) | 47 | 68
mg/dL | 7.9124 [-0.6975 to 16.5224] | -1.6217 [-9.2467 to 6.0033]

14. Secondary Outcome: Change in Systolic Blood Pressure (Stage 2: Usual Care v. Mentee)
Description: as for outcome 5
Time Frame: Baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: mmHG
Arm/Group | Stage 2 Usual Care | Stage 2 Peer Mentoring FFM (From Former Mentee)
Number analyzed (Participants) | 47 | 68
mmHG | 1.4718 [-3.5255 to 6.4692] | 0.1876 [-4.0493 to 4.4244]

15. Secondary Outcome: Change in Diabetes Quality of Life (Stage 2: Usual Care v. Mentee)
Description: as for outcome 6
Time Frame: Baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stage 2 Usual Care | Stage 2 Peer Mentoring FFM (From Former Mentee)
Number analyzed (Participants) | 47 | 68
score on a scale | 0.1024 [-0.2040 to 0.4089] | -0.4098 [-0.6816 to -0.1380]

16. Secondary Outcome: Change in Depression Symptoms (Stage 2: Usual Care v. Mentees)
Description: as for outcome 7
Time Frame: Baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stage 2 Usual Care | Stage 2 Peer Mentoring FFM (From Former Mentee)
Number analyzed (Participants) | 47 | 68
score on a scale | -0.3186 [-0.7744 to 0.1373] | -0.2627 [-0.6723 to 0.1469]

17. Secondary Outcome: Change in Glucose Control (Stage 2: Usual Care v. Mentees)
Description: as for outcome 8
Time Frame: Baseline to 12 months
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Stage 2 Usual Care | Stage 2 Peer Mentoring FFM (From Former Mentee)
Number analyzed (Participants) | 47 | 68
percent | -0.2661 [-0.8889 to 0.3567] | -0.1628 [-0.6544 to 0.3287]

18. Secondary Outcome: Change in Direct LDL Blood Levels (Stage 2: Usual Care v. Mentees)
Description: as for outcome 9
Time Frame: Baseline to 12 months
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Stage 2 Usual Care | Stage 2 Peer Mentoring FFM (From Former Mentee)
Number analyzed (Participants) | 47 | 68
mg/dL | 5.0419 [-4.0961 to 14.1799] | -4.9126 [-12.8131 to 2.9879]

19. Secondary Outcome: Change in Systolic Blood Pressure (Stage 2: Usual Care v. Mentee)
Description: as for outcome 10
Time Frame: Baseline to 12 months
Measure: Mean (95% Confidence Interval); unit: mmHG
Arm/Group | Stage 2 Usual Care | Stage 2 Peer Mentoring FFM (From Former Mentee)
Number analyzed (Participants) | 47 | 68
mmHG | -1.6851 [-6.8849 to 3.5147] | 1.3877 [-2.7712 to 5.5466]

20. Secondary Outcome: Change in Diabetes Quality of Life (Stage 2: Usual Care v. Mentee)
Description: as for outcome 11
Time Frame: Baseline to 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stage 2 Usual Care | Stage 2 Peer Mentoring FFM (From Former Mentee)
Number analyzed (Participants) | 47 | 68
score on a scale | -0.1299 [-0.4464 to 0.1866] | -0.0246 [-0.3058 to 0.2567]

21. Secondary Outcome: Change in Depression Symptoms (Stage 2: Usual Care v. Mentees)
Description: as for outcome 12
Time Frame: Baseline to 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stage 2 Usual Care | Stage 2 Peer Mentoring FFM (From Former Mentee)
Number analyzed (Participants) | 47 | 68
score on a scale | -0.4581 [-0.9375 to 0.0214] | -0.0890 [-0.5157 to 0.3377]

22. Secondary Outcome: Change in Direct LDL Blood Levels (Stage 2: Non-mentors v. Mentors)
Description: as for outcome 4
Time Frame: Baseline to 6 months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Stage 2 Non-mentor | Stage 2 Mentor
Number analyzed (Participants) | 69 | 70
mg/dL | -2.1692 [-9.0874 to 4.7491] | -7.4649 [-14.2567 to -0.6732]

23. Secondary Outcome: Change in Systolic Blood Pressure (Stage 2: Non-mentors v. Mentors)
Description: as for outcome 5
Time Frame: Baseline to 6 months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: mmHG
Arm/Group | Stage 2 Non-mentor | Stage 2 Mentor
Number analyzed (Participants) | 69 | 70
mmHG | -1.6942 [-5.6326 to 2.2443] | -1.0527 [-5.2420 to 3.1366]

24. Secondary Outcome: Change in Diabetes Quality of Life (Stage 2: Non-mentors v. Mentors)
Description: as for outcome 6
Time Frame: Baseline to 6 months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stage 2 Non-mentor | Stage 2 Mentor
Number analyzed (Participants) | 69 | 70
score on a scale | -0.1006 [-0.3213 to 0.1202] | -0.1332 [-0.3574 to 0.0910]

25. Secondary Outcome: Change in Depression Symptoms (Stage 2: Non-mentors v. Mentors)
Description: as for outcome 7
Time Frame: Baseline to 6 months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stage 2 Non-mentor | Stage 2 Mentor
Number analyzed (Participants) | 69 | 70
score on a scale | -0.3314 [-0.6916 to 0.0288] | -0.1809 [-0.5454 to 0.1837]

26. Secondary Outcome: Change in Glucose Control (Stage 2: Non-mentors v. Mentors)
Description: as for outcome 8
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Stage 2 Non-mentor | Stage 2 Mentor
Number analyzed (Participants) | 69 | 70
percent | 0.2396 [-0.1853 to 0.6645] | 0.0639 [-0.3306 to 0.4585]

27. Secondary Outcome: Change in Direct LDL Blood Levels (Stage 2: Non-mentors v. Mentors)
Description: as for outcome 9
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Stage 2 Non-mentor | Stage 2 Mentor
Number analyzed (Participants) | 69 | 70
mg/dL | -1.0938 [-8.3514 to 6.1637] | 2.2494 [-4.7631 to 9.2619]

28. Secondary Outcome: Change in Systolic Blood Pressure (Stage 2: Non-mentors v. Mentors)
Description: as for outcome 10
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: mmHG
Arm/Group | Stage 2 Non-mentor | Stage 2 Mentor
Number analyzed (Participants) | 69 | 70
mmHG | -3.9453 [-8.1308 to 0.2401] | -0.5611 [-4.7598 to 3.6375]

29. Secondary Outcome: Change in Diabetes Quality of Life (Stage 2: Non-mentors v. Mentors)
Description: as for outcome 11
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stage 2 Non-mentor | Stage 2 Mentor
Number analyzed (Participants) | 69 | 70
score on a scale | -0.1896 [-0.4311 to 0.0519] | -0.3017 [-0.5475 to -0.0559]

30. Secondary Outcome: Change in Depression Symptoms (Stage 2: Non-mentors v. Mentors)
Description: as for outcome 12
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stage 2 Non-mentor | Stage 2 Mentor
Number analyzed (Participants) | 69 | 70
score on a scale | 0.0609 [-0.3251 to 0.4470] | -0.0819 [-0.4716 to 0.3077]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 18 months from baseline.
Groups:
- Usual Care Stage 1; Usual Care Stage 2: No interventions will be provided to this arm. They will complete planned surveys, and blood draws (baseline, 6 months, and 12 months).
Arm/Group | Usual Care Stage 1 | Peer Mentoring | Peer Mentoring FFM (From Former Mentee) | Usual Care Stage 2
All-Cause Mortality (participants affected / at risk) | 2/156 | 3/205 | 2/70 | 2/49
Serious Adverse Events (participants affected / at risk) | 10/156 | 28/205 | 12/70 | 2/49
Other Adverse Events (participants affected / at risk) | 11/156 | 38/205 | 6/70 | 5/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care Stage 1 (N=156) | Peer Mentoring (N=205) | Peer Mentoring FFM (From Former Mentee) (N=70) | Usual Care Stage 2 (N=49)
Hospitalization (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2) | 0 (0) — We considered any hospitalization (any participant who had to stay in the hospital overnight due to their condition) an SAE. Therefore, these numbers represent those who were hospitalized as a result of an SAE.
Hospitalization (General disorders) | 4 (4) | 15 (15) | 3 (4) | 1 (1) — We considered any hospitalization (any participant who had to stay in the hospital overnight due to their condition) an SAE. Therefore, these numbers represent those who were hospitalized as a result of an SAE.
Hospitalization (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 0 (0) — We considered any hospitalization (any participant who had to stay in the hospital overnight due to their condition) an SAE. Therefore, these numbers represent those who were hospitalized as a result of an SAE.
Hospitalization (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — We considered any hospitalization (any participant who had to stay in the hospital overnight due to their condition) an SAE. Therefore, these numbers represent those who were hospitalized as a result of an SAE.
Hospitalization (Renal and urinary disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0) — We considered any hospitalization (any participant who had to stay in the hospital overnight due to their condition) an SAE. Therefore, these numbers represent those who were hospitalized as a result of an SAE.
Hospitalization (Surgical and medical procedures) | 1 (1) | 2 (2) | 1 (1) | 1 (1) — We considered any hospitalization (any participant who had to stay in the hospital overnight due to their condition) an SAE. Therefore, these numbers represent those who were hospitalized as a result of an SAE.
Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (3) | 1 (1) — We considered any hospitalization (any participant who had to stay in the hospital overnight due to their condition) an SAE. Therefore, these numbers represent those who were hospitalized as a result of an SAE.
Hospitalization (Immune system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) — We considered any hospitalization (any participant who had to stay in the hospital overnight due to their condition) an SAE. Therefore, these numbers represent those who were hospitalized as a result of an SAE.
Hospitalization (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — We considered any hospitalization (any participant who had to stay in the hospital overnight due to their condition) an SAE. Therefore, these numbers represent those who were hospitalized as a result of an SAE.
Hospitalization (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — We considered any hospitalization (any participant who had to stay in the hospital overnight due to their condition) an SAE. Therefore, these numbers represent those who were hospitalized as a result of an SAE.
Hospitalization (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — We considered any hospitalization (any participant who had to stay in the hospital overnight due to their condition) an SAE. Therefore, these numbers represent those who were hospitalized as a result of an SAE.
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — We considered any hospitalization (any participant who had to stay in the hospital overnight due to their condition) an SAE. Therefore, these numbers represent those who were hospitalized as a result of an SAE.
Hospitalization (Cardiac disorders) | 0 (0) | 6 (8) | 5 (9) | 1 (1) — We considered any hospitalization (any participant who had to stay in the hospital overnight due to their condition) an SAE. Therefore, these numbers represent those who were hospitalized as a result of an SAE.
Hospitalization (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — We considered any hospitalization (any participant who had to stay in the hospital overnight due to their condition) an SAE. Therefore, these numbers represent those who were hospitalized as a result of an SAE.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care Stage 1 (N=156) | Peer Mentoring (N=205) | Peer Mentoring FFM (From Former Mentee) (N=70) | Usual Care Stage 2 (N=49)
ED visit (Injury, poisoning and procedural complications) | 3 (3) | 7 (8) | 3 (3) | 1 (1) — We considered any ED visit (any participant who went to the emergency room due to their condition) an AE. Therefore, these numbers represent those who went to the emergency room as a result of an AE.
ED visit (Surgical and medical procedures) | 3 (3) | 4 (6) | 2 (2) | 2 (2) — We considered any ED visit (any participant who went to the emergency room due to their condition) an AE. Therefore, these numbers represent those who went to the emergency room as a result of an AE.
ED visit (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — We considered any ED visit (any participant who went to the emergency room due to their condition) an AE. Therefore, these numbers represent those who went to the emergency room as a result of an AE.
ED visit (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — We considered any ED visit (any participant who went to the emergency room due to their condition) an AE. Therefore, these numbers represent those who went to the emergency room as a result of an AE.
ED visit (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) — We considered any ED visit (any participant who went to the emergency room due to their condition) an AE. Therefore, these numbers represent those who went to the emergency room as a result of an AE.
ED visit (General disorders) | 1 (1) | 21 (26) | 0 (0) | 2 (2) — We considered any ED visit (any participant who went to the emergency room due to their condition) an AE. Therefore, these numbers represent those who went to the emergency room as a result of an AE.
ED visit (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — We considered any ED visit (any participant who went to the emergency room due to their condition) an AE. Therefore, these numbers represent those who went to the emergency room as a result of an AE.
ED visit (Infections and infestations) | 0 (0) | 4 (5) | 0 (0) | 1 (1) — We considered any ED visit (any participant who went to the emergency room due to their condition) an AE. Therefore, these numbers represent those who went to the emergency room as a result of an AE.
ED visit (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5) | 1 (1) | 0 (0) — We considered any ED visit (any participant who went to the emergency room due to their condition) an AE. Therefore, these numbers represent those who went to the emergency room as a result of an AE.
ED visit (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — We considered any ED visit (any participant who went to the emergency room due to their condition) an AE. Therefore, these numbers represent those who went to the emergency room as a result of an AE.
ED visit (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — We considered any ED visit (any participant who went to the emergency room due to their condition) an AE. Therefore, these numbers represent those who went to the emergency room as a result of an AE.
ED visit (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — We considered any ED visit (any participant who went to the emergency room due to their condition) an AE. Therefore, these numbers represent those who went to the emergency room as a result of an AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT01651117/Prot_SAP_000.pdf